CLINICAL TRIAL: NCT03824561
Title: Special Drug-Use Surveillance Study on Entyvio for IV Infusion 300 mg [Ulcerative Colitis]
Brief Title: Special Drug-Use Surveillance Study on Vedolizumab for IV Infusion 300 mg [Ulcerative Colitis]
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-5033; jRCT1080224534 (Registry Identifier: jRCT)
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab; Infusions, Intravenous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vedolizumab 300 mg: Vedolizumab IV infusion 300 mg, at Weeks 0, 2 and 6, and every 8 weeks thereafter, for up to 54 weeks. Participants will receive IV infusion as part of routine medical care.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab IV infusion
  Other Names: Entyvio for IV Infusion 300 mg

SUMMARY:
The purpose of this survey is to evaluate the long-term safety and effectiveness of vedolizumab for intravenous (IV) infusion 300 milligrams (mg) in ulcerative colitis (UC) patients in the routine clinical setting.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab for IV infusion 300 mg. This drug is being tested to treat patients who have UC.

This study is an observational (non-interventional) study and will look at the long-term safety and effectiveness of vedolizumab for IV infusion 300 mg in the routine clinical setting. The planned number of observed patients will be approximately 1,000.

This multi-center observational trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Have moderate or severe active UC
2. Have inadequate response to existing therapies

Exclusion Criteria:

Patients with any contraindication for vedolizumab

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: UC patients treated with vedolizumab for IV infusion 300 mg as part of routine medical care
Sampling Method: Non-Probability Sample
Enrollment: 1110 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Matsuoka K, Hisamatsu T, Mikami Y, Yamamoto T, Motoya S, Shinzaki S, Iwakiri R, Sugiura K, Nishimura K, Kajita M, Fernandez JL. Safety and Effectiveness of Vedolizumab in Patients with Moderate-to-Severe Ulcerative Colitis: An Interim Analysis of a Japanese Post-Marketing Surveillance Study. Adv Ther. 2023 Jun;40(6):2902-2914. doi: 10.1007/s12325-023-02500-6. Epub 2023 May 4. PMID 37140705
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b603a4db2bf003ab4a2c9

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 197 investigative sites in Japan, from 1 February 2019 to 12 February 2025.
Pre-assignment Details: Participants with ulcerative colitis who received Vedolizumab IV infusion 300 mg were enrolled. Participants received Vedolizumab IV infusion 300 mg as part of a routine normal practice.
Groups:
- Vedolizumab 300 mg: Vedolizumab IV infusion 300 mg, at Weeks 0, 2 and 6, and every 8 weeks thereafter, for up to 54 weeks. Participants received IV infusion as part of routine normal practice.
Period: Overall Study
Arm/Group | Vedolizumab 300 mg
Started | 1110
Completed | 1091
Not Completed | 19
Not completed — Protocol Violation | 19

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the study.
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 1091
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (17.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 470
  Male | 621
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Events (AEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not the event is considered causally related to the use of the product.
Time Frame: Up to Week 54
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 1091
Participants | 208

2. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Drug Reactions
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not the event is considered causally related to the use of the product. Adverse drug reaction refers to AE related to administered drug.
Time Frame: Up to Week 54
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 1091
Participants | 60

3. Secondary Outcome: Number of Participants Who Had a Presence or Absence of Therapeutic Response After 3 Doses of Vedolizumab
Time Frame: Week 54
Population: Efficacy analysis set: The efficacy analysis set was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available.
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 1062
Participants
  With Presence | 904
  With Absence | 158

4. Secondary Outcome: Number of Participants Who Continued the Therapy After 3 Doses of Vedolizumab
Time Frame: Week 54
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 1062
Participants
  Continued Participants | 880
  Not Continued Participants | 182

5. Secondary Outcome: Change From Baseline in Complete Mayo Scores
Description: Mayo score is used to assess UC disease activity. It consists of 4 sub-scores (stool frequency, rectal bleeding, findings on sigmoidoscopy, and physician's global assessment), each ranges from 0 to 3. Complete Mayo score sums 4 subscores and ranges from 0 to 12, with higher scores indicating more severe disease.
Time Frame: Baseline and Week 54
Population: Efficacy analysis set: The efficacy analysis set was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. The analyzed numbers were participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 32
score on a scale | -2.1 (3.67)

6. Secondary Outcome: Change From Baseline in Partial Mayo Scores
Description: Mayo score is used to assess UC disease activity. It consists of 4 sub-scores (stool frequency, rectal bleeding, findings on sigmoidoscopy, and physician's global assessment), each ranges from 0 to 3. Partial Mayo score sums 3 subscores excluding the sigmoidoscopy sub-score and ranges from 0 to 9, with higher scores indicating more severe disease.
Time Frame: Baseline and Week 54
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 590
score on a scale | -3.4 (2.42)

7. Secondary Outcome: Change From Baseline in Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Score
Description: The SIBDQ is an instrument used to assess quality of life (QOL) and is a disease-specific health-related quality of life questionnaire, that consists of 10 questions, each question is scored on a scale from 1 (poor quality of life) to 7 (good quality of life). The total score is ranging from 10 to 70 with a higher score indicates a better health-related quality of life. Change from Baseline in SIBDQ total score was reported.
Time Frame: Baseline and Week 54
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 653
score on a scale | 9.3 (12.86)

ADVERSE EVENTS:
Time Frame: Up to Week 54
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the study treatment.
Arm/Group | Vedolizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 5/1091
Serious Adverse Events (participants affected / at risk) | 82/1091
Other Adverse Events (participants affected / at risk) | 29/1091
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 300 mg (N=1091)
Appendicitis (Infections and infestations) | 3
Atypical pneumonia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis Escherichia coli (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Cytomegalovirus enterocolitis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Herpes zoster oticus (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Cerebral infarction (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 37
Haematochezia (Gastrointestinal disorders) | 1
Intussusception (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Pancreatitis acute (Gastrointestinal disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Paroxysmal nocturnal haemoglobinuria (Renal and urinary disorders) | 1
Diabetic nephropathy (Renal and urinary disorders) | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1
Pyrexia (General disorders) | 1
Neutrophil toxic granulation present (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 300 mg (N=1091)
Nasopharyngitis (Infections and infestations) | 15
Infusion related reaction (Injury, poisoning and procedural complications) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT03824561/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT03824561/SAP_001.pdf